CLINICAL TRIAL: NCT05444634
Title: The Effect of Distraction Cards and Stress Ball on Pain and Anxiety in Children With Intramuscular Injection
Brief Title: The Pain and Anxiety in Children With Intramuscular Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Collaborators: MSc Merve Eroğlu (Unknown)
Responsible Party: Principal Investigator, Türkan Kadiroğlu, Director, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.O.01.00/265
Record Dates: First submitted 2022-04-29; First posted 2022-07-06 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Intramuscular Myxoma
Keywords: Children; Pain, Acute; Anxiety
MeSH Terms: conditions — Acute Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- distraction card (Experimental): Immediately before the procedure, the child will be asked questions about the distraction cards. Questions about the cards will continue to be asked immediately after the intramuscular injection is finished.
  Interventions: Behavioral: Distraction Card
- Stress Ball (Experimental): The child will be informed about the stress ball and asked to play continuously
  Interventions: Behavioral: Stress Ball
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Distraction Card — Suitable for children over 3 years old. 1 set of 32 pieces of thick cardboard cards It has been prepared by child development experts in line with pedagogical principles.
  Size: 13cm x 8cm, Each card illustrates the skills and actions the children do.
  Arms: distraction card
Behavioral: Stress Ball — Brain Shaped Stress Ball, White rope in the form of mesh around the inner silicone Size: Approx 2.4 inches (6 cm), Color: Colorful, When squeezed, the silicone structure comes out in the mesh spaces and turns into a bunch of grapes.
  Arms: Stress Ball

SUMMARY:
This study was planned as a randomized controlled experimental study to determine the effect of distraction cards and stress ball on pain and anxiety in children with intramuscular injection.

DETAILED DESCRIPTION:
Pharmacological and non-pharmacological methods are used in the management of pain and anxiety in children. Non-pharmacological methods are noninvasive, inexpensive, have no side effects and are independent functions of the nurse.This study was planned as a randomized controlled experimental study to determine the effect of distraction cards and stress ball on pain and anxiety in children with intramuscular injection. The study was conducted between May 2022 and August 2022. It will be done with children aged 3-6 years who come to the emergency unit of the State Hospital, who are given intramuscular injection.

"Descriptive Information Form", "Wong Baker Faces Pain Rating Scale", "Venham Anxiety Rating Picture Scale" will be used in data collection.

ELIGIBILITY:
Inclusion Criteria:

* 3-6 years old
* Intramuscular administration of ondansetron hcl active ingredient drug
* Mentally and physically handicapped
* Does not have a disease that causes chronic pain
* Open to communication
* Fluent in Turkish

Exclusion Criteria:

* Children of parents who did not give written consent
* Children who do not give verbal consent appropriate to the child's developmental level

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Pain, acute | 12 week
  Wong Baker Faces Pain Rating Scale:
  This scale was developed by Donna Wong and Connie Morain Baker in 1981 and later revised in 1983.
  The scale is suitable for describing the pain status of children aged 3-18 years.
  Children can express many pain areas and their severity with this scale. There are 6 facial expressions in the scale. The scores of "0", "2", "4", "6", "8", "10" were indicated for each facial expression, respectively.
  Facial expressions are given points with the lowest "0" and the highest "10". A score of "0" was defined as no pain, while a score of "10" was defined as unbearable pain.
Anxiety, spitefulness | 12 week
  Venham Anxiety Rating Picture Scale:
  The scale was developed by Larry L. Venham and Elise Gaulin Kremer in 1979. The scale is used to determine the anxiety status of children over 3 years old. There are 8 cards in the scale and two pictures on each card. Cards 1 to 8 are shown to the child in turn.
  Of the pictures, the anxious picture is given 1 point, while the non-anxious picture is given 0 points.
  The lowest is 0 points, while the highest is 8 points. In the 0 to 8 scoring system, the higher the score, the higher the anxiety rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Erzuum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No